CLINICAL TRIAL: NCT04959968
Title: The Effect of Use of Eye Bands and Earplugs on Sleep Quality, Anxiety and Comfort Level in Patients Undergoing Craniotomy Surgery
Brief Title: The Use of Eye Patches and Earplugs in Intensive Care in Cases of Craniotomy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taksim Egitim ve Arastirma Hastanesi (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TaksimEğitim
Record Dates: First submitted 2021-06-25; First posted 2021-07-13 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2022-10

CONDITIONS: Craniotomy
Keywords: Anxiety; Sleep; Intensive Care, Surgical; Craniotomy
MeSH Terms: conditions — Anxiety Disorders | interventions — Ear Protective Devices

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): An eye patch and earplug will be applied to the intervention group in the intensive care unit on the day of craniotomy and on the post-operative 1st day between 22:00 and 06:00
  Interventions: Device: eye patch and earplug
- Control group (No Intervention): Standard care procedure will be applied to the control group

INTERVENTIONS:
Device: eye patch and earplug — The use of eye patch and ear plugs in post-operative intensive care in craniotomy cases.
  Arms: Intervention group

SUMMARY:
This study aims to evaluate the effects of using eye patch and earplugs on anxiety, patient comfort, and sleep quality after craniotomy. The study will be carried out in a hospital located in the Northwest of Turkey. A total of 60 patients meeting the research criteria will be randomized to intervention and control groups. An eye patch and earplug will be applied to the intervention group in the intensive care unit on the day of craniotomy and on the post-operative 1st day between 22:00 and 06:00. Standard care procedure will be applied to the control group. Richard-Campbell Sleep Questionnaire, Aktiwatch, Hospital Anxiety and Depression Scale and General Comfort Questionnaire will be used to collect study data.

DETAILED DESCRIPTION:
This study was designed as a non-drug clinical study with 2 randomly selected groups to evaluate the effect of eye patch and earplug use on sleep quality, anxiety and comfort level in patients hospitalized in the intensive care unit after craniotomy. The study will be carried out in a hospital located in the Northwest of Turkey. A total of 60 patients meeting the research criteria will be randomized to intervention and control groups. An eye patch and earplug will be applied to the intervention group in the intensive care unit on the day of craniotomy and on the post-operative 1st day between 22:00 and 06:00. Standard care procedure will be applied to the control group. Richard-Campbell Sleep Questionnaire, Aktiwatch, Hospital Anxiety and Depression Scale and General Comfort Questionnaire will be used to collect study data.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective craniotomy and intensive care for at least 48 hours
* Glasgow Coma Scale score = 15
* Turkish literate

Exclusion Criteria:

* Diagnosis of sleep disorder
* Hearing and/or vision loss
* Hearing aid use
* Pregnant women
* Communication and/or cooperation problem
* Chronic pain medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-10 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-06-17 (Actual)

PRIMARY OUTCOMES:
The Richards-Campbell Sleep Questionnaire | On the 1 day of craniotomy
  Sleep quality levels of the craniotomy cases
The Richards-Campbell Sleep Questionnaire | Post-operative second day of craniotomy
  Sleep quality levels of the craniotomy cases

SECONDARY OUTCOMES:
The Hospital Anxiety and Depression Scale | On the 1 day of craniotomy
  Anxiety levels of the craniotomy cases
The Hospital Anxiety and Depression Scale | Post-operative second day of craniotomy
  Anxiety levels of the craniotomy cases
The General Comfort Questionnaire | Post-operative second day of craniotomy
  General comfort levels of the craniotomy cases

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpaşa Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No